CLINICAL TRIAL: NCT01337258
Title: Economic Analyses Alongside the REDUCE Clinical Trial
Brief Title: Economic Analyses of the REDUCE Trial
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113979
Record Dates: First submitted 2010-03-04; First posted 2011-04-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms, Prostate; Benign Prostatic Hyperplasia; Cancer
Keywords: cost effectiveness; dutasteride; elevated risk population; Prostate cancer; prevention
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia; Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men at increased risk for Prostate Cancer (PCA)
  Interventions: Drug: Dutasteride; Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — dutasteride 0.5mg daily.
  Other Names: Placebo
Drug: Placebo — Men taking placebo daily

SUMMARY:
The objective of this project is to conduct a retrospective economic analysis of the use of dutasteride for the prevention of prostate cancer based on data from the REDUCE clinical trial. REDUCE is a 4-year, phase 3, randomized, double-blind, parallel assignment clinical trial of the use of dutasteride compared with no chemopreventive treatment.

The REDUCE trial was a four-year, international, multicenter, randomized, double-blind, placebo-controlled, parallel group study. There were 790 investigators in 42 countries.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 50 to 75 years
* serum prostate-specific antigen (PSA) ≥2.5 ng per milliliter and ≤10 ng per milliliter (men aged 50-60 years) or ≥3.0 ng per milliliter and ≤10 ng per milliliter (men aged >60 years)
* single, negative prostate biopsy (6-12 cores) within 6 months prior to enrollment (independent of the study)

Exclusion Criteria:

* Principal exclusion criteria were more than one prior prostate biopsy
* high-grade intraepithelial neoplasia (HG-PIN) or atypical small acinar proliferation (ASAP) on the pre-entry prostate biopsy
* a prostate volume >80 ml, previous prostate surgery
* International Prostate Symptom Score (IPSS) ≥25 or ≥20 if already on alpha-blocker therapy for BPH

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men at increase risk for prostate cancer ages 50-75 who were enrolled in the REDUCE study
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cost of treating prostate-related events | REDUCE clinical trial, 4 year time period
  Prostate Related Events include Benign Prostatic Hyperplasia (BPH), Prostate Cancer (PCA) and Prostatitis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline